CLINICAL TRIAL: NCT05543252
Title: A Dose-Blinded Extension Study to Evaluate the Long-Term Efficacy, Safety, and Tolerability of UCB0599 in Study Participants With Parkinson's Disease
Brief Title: An Extension Study to Evaluate the Long-Term Efficacy, Safety and Tolerability of Minzasolmin (UCB0599) in Study Participants With Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on available data, the decision was made to stop development of UCB0599/minzasolmin as treatment of Parkinson's Disease.
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PD0055; 2022-500424-30-00 (Registry Identifier: EU CT Number); U1111-1279-2323 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease.; UCB0599; Phase 2; Minzasolmin
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minzasolmin (UCB0599) High Dose Arm (Experimental): Participants will receive a predefined high dosage of minzasolmin (UCB0599) during the Treatment Period.
  Interventions: Drug: Minzasolmin (UCB0599)
- Minzasolmin (UCB0599) Low Dose Arm (Experimental): Participants will receive a predefined low dosage of minzasolmin (UCB0599) during the Treatment Period.
  Interventions: Drug: Minzasolmin (UCB0599)

INTERVENTIONS:
Drug: Minzasolmin (UCB0599) — Minzasolmin (UCB0599) Pharmaceutical form: Granules in capsules Route of administration: Oral use Participants will receive minzasolmin (UCB0599) in a pre-specified sequence during the Treatment Period.

SUMMARY:
The purpose of the study is to estimate the pharmacodynamic effects of minzasolmin (UCB0599) on brain pathophysiology in Early-start versus Delayed-start participants originally diagnosed with new onset Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria

* Participant completed the Treatment Period of PD0053 (NCT04658186). The Baseline Visit for PD0055 (Visit 2) should be no later than 4 weeks following the end of treatment (EOT) Visit in PD0053 (NCT04658186). Any delay needs to be justified by the Investigator and approved by the Sponsor
* A male study participant must agree to use contraception during the Treatment Period and for at least 90 days after the last dose of the IMP and refrain from donating sperm during this period.
* A female study participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  ◦ Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 1 month after the last dose of investigational medicinal product (IMP). The study participant must have a negative urine pregnancy test at Screening (Visit 1), which is to be confirmed negative by urine testing prior to the first dose of IMP at PD0055 Baseline Visit. If oral contraception is used, an additional barrier method will be required during the study as an IMP-related gastrointestinal upset or a drug interaction by cytochrome P450 3A4 (CYP3A4) induction could interfere with efficacy
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent form (ICF) and in this protocol.

Exclusion Criteria:

* Study participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* A female study participant who tests positive for pregnancy, plans to get pregnant during the participation in the study, or who is breastfeeding
* Study participant had previously participated in PD0055
* Study participant meets any withdrawal criteria in PD0053 (NCT04658186)
* Study participants wearing any kind of implantable active device, including cardiac pacemakers, pumps, and implantable cardioverters, will be excluded from using Digital Health Technology, but may participate in the main study
* Study participant does not agree to refrain from donating blood or blood products or other body fluids

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Baseline adjusted Dopamine Transporter Imaging with Single Photon Emission Computed Tomography (DaT-SPECT) whole striatum SBR at PD0055 Month 18 | From Baseline up to Month 18
  The change from baseline (screening) in mean striatum specific binding ratios (SBR) will be assessed by Dopamine Transporter Imaging with Single Photon Emission Computed Tomography using 123I-Ioflupane as radiopharmaceutical.
  Baseline will refer to PD0053 (NCT04658186) Screening Visit date.

SECONDARY OUTCOMES:
Cumulative Levodopa Equivalent Daily Dose; (LEDD) at PD0055 Month 18 | From Baseline up to Month 18
  The Cumulative Levodopa Equivalent Daily Dose (LEDD) will be calculated for each participant at each visit and at the end of study. This is the sum of all the LEDDs taken up to that visit. Any changes in medication (type, dose, or dosing regimen) should be accounted for when calculating cumulative doses.
Incidence of treatment-emergent adverse event (TEAEs) | From Baseline to the Safety Follow-up Visit (Month 31)
  Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Incidence of serious adverse events (SAEs) | From Baseline to the Safety Follow-up Visit (Month 31)
  Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Serious criteria of death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect . Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Incidence of TEAEs leading to withdrawal from study | From Baseline to the Safety Follow-up Visit (Month 31)
  Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (96):
- United States (41):
  - Pd0055 50506, Phoenix, Arizona
  - Pd0055 50519, Fountain Valley, California
  - Pd0055 50385, Fresno, California
  - Pd0055 50118, Los Angeles, California
  - Pd0055 50531, Englewood, Colorado
  - Pd0055 50392, Danbury, Connecticut
  - Pd0055 50538, Farmington, Connecticut
  - Pd0055 50396, Boca Raton, Florida
  - Pd0055 50524, Bradenton, Florida
  - Pd0055 50394, Tampa, Florida
  - Pd0055 50544, Augusta, Georgia
  - Pd0055 50401, Chicago, Illinois
  - Pd0055 50310, Chicago, Illinois
  - Pd0055 50399, Winfield, Illinois
  - Pd0055 50549, Iowa City, Iowa
  - Pd0055 50074, Kansas City, Kansas
  - Pd0055 50121, Lexington, Kentucky
  - Pd0055 50395, New Orleans, Louisiana
  - Pd0055 50547, Baltimore, Maryland
  - Pd0055 50243, Boston, Massachusetts
  - Pd0055 50546, Worcester, Massachusetts
  - Pd0055 50386, Farmington Hills, Michigan
  - Pd0055 50536, Saint Paul, Minnesota
  - Pd0055 50397, Las Vegas, Nevada
  - Pd0055 50530, Stony Brook, New York
  - Pd0055 50535, Williamsville, New York
  - Pd0055 50372, Cleveland, Ohio
  - Pd0055 50311, Cleveland, Ohio
  - Pd0055 50255, Columbus, Ohio
  - Pd0055 50398, Tulsa, Oklahoma
  - Pd0055 50084, Charleston, Oregon
  - Pd0055 50526, Philadelphia, Pennsylvania
  - Pd0055 50543, Memphis, Tennessee
  - Pd0055 50113, Houston, Texas
  - Pd0055 50525, Houston, Texas
  - Pd0055 50400, San Antonio, Texas
  - Pd0055 50107, Burlington, Vermont
  - Pd0055 50410, Fairfax, Virginia
  - Pd0055 50534, Virginia Beach, Virginia
  - Pd0055 50292, Kirkland, Washington
  - Pd0055 50402, Crab Orchard, West Virginia
- Canada (3):
  - Pd0055 50374, Calgary
  - Pd0055 50387, Ottawa
  - Pd0055 50389, Toronto
- France (9):
  - Pd0055 40527, Bordeaux
  - Pd0055 40424, Créteil
  - Pd0055 40526, Lille
  - Pd0055 40130, Marseille
  - Pd0055 40635, Nantes
  - Pd0055 40524, Nîmes
  - Pd0055 40525, Paris
  - Pd0055 40131, Strasbourg
  - Pd0055 40528, Toulouse
- Germany (11):
  - Pd0055 40515, Berlin
  - Pd0055 40138, Bonn
  - Pd0055 40530, Dresden
  - Pd0055 40711, Erbach im Odenwald
  - Pd0055 40023, Erlangen
  - Pd0055 40710, Essen
  - Pd0055 40532, Haag in Oberbayern
  - Pd0055 40249, Kiel
  - Pd0055 40174, Mainz
  - Pd0055 40529, Marburg
  - Pd0055 40531, Regensburg
- Italy (5):
  - Pd0055 40555, Brescia
  - Pd0055 40533, Padua
  - Pd0055 40257, Roma
  - Pd0055 40534, Roma
  - Pd0055 40697, Terni
- Pd0055 40359, Nijmegen, Netherlands
- Poland (11):
  - Pd0055 40694, Bydgoszcz
  - Pd0055 40719, Jelenia Góra
  - Pd0055 40539, Katowice
  - Pd0055 40538, Krakow
  - Pd0055 40696, Krakow
  - Pd0055 40700, Lodz
  - Pd0055 40702, Lublin
  - Pd0055 40535, Oświęcim
  - Pd0055 40536, Warsaw
  - Pd0055 40699, Warsaw
  - Pd0055 40705, Warsaw
- Spain (9):
  - Pd0055 40045, A Coruña
  - Pd0055 40159, Barcelona
  - Pd0055 40267, Barcelona
  - Pd0055 40046, Córdoba
  - Pd0055 40540, Madrid
  - Pd0055 40542, Móstoles
  - Pd0055 40352, Pamplona
  - Pd0055 40541, San Sebastián
  - Pd0055 40049, Seville
- United Kingdom (6):
  - Pd0055 40175, London
  - Pd0055 40543, London
  - Pd0055 40698, London
  - Pd0055 40544, Motherwell
  - Pd0055 40306, Newcastle upon Tyne
  - Pd0055 40457, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/